CLINICAL TRIAL: NCT05565651
Title: Retrospective Study for the Characterization of the Intestinal Microbiota in Association With Pathologies and Diet in the Italian Population
Brief Title: Retrospective Study of Intestinal Microbiota in Association With Diabetes
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, FRANCESCA DI GAUDIO, Researcher, University of Palermo
Other Study IDs: 8/14/2022
Record Dates: First submitted 2022-09-23; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Dysbiosis Symptoms Linked to Pathology
Keywords: Microbiote; Dysbiosis
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fecal microbiota analysis — Data analysis

SUMMARY:
The microbiota interacts with several human organs and influences the physiological process in the host. The predominant Phyla of species in the gut microbiota are Bacteroidetes (B) and Firmicutes (F), accounting for 60-80%, and Proteobacteria (P) and Actinobacteria (A) in minority. When some of the bacterial Phyla species are unbalanced, the pathological state of dysbiosis occurs. A laboratory index used for clinical analyzes is the F / B ratio <0.8, which characterizes an intestinal dysbiotic state.

Many causes can affect the intestinal microbiota, thus altering it in a dysbiotic state, first of all the diet. In fact, dysbiosis can be characterized both by the severity with which it manifests itself and is also distinguished in putrefactive and fermentative dysbiosis.

Furthermore, the variation in the "normal" percentages of the Phyla is also related to some pathological alterations.

The aim of this study will be to monitor the population and heterogeneity of the microbiota in the Italian population. Knowing the complex implications of dysbiosis and the extensive data on it, this study will want to detail the state of the gut microbiota in the previously indicated population, focusing attention on peculiar profiles that could reflect a pathogenic spectrum or metabolic disturbances.

The study aims to investigate the diffusion and state of the microbiota in the Italian territory and if it occurs in association with certain pathologies and / or diet.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 16 and 80 years old,
* Patients with completed questionnare
* Dysbiosis symptoms

Exclusion Criteria:

* Under 16 years old,
* over 80 years old,
* patients misidentified

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male and Female
Study Population: 334 fecal samples from Lifebrain Cerba Healthcare Italian laboratory network were analyzed to perform a gut microbiota genetic test, accompanied by filling an attachment to provide a medical history useful for the interpretation of the results obtained and to provide a correct diagnosis using a specific test kit for the stool sample collection. The samples were collected from people aged between 2 and 87 years old.
Sampling Method: Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Outcome percentage Phyla | 2020-2022
  Change in the percentage of Proteobacteria in type 2 diabetic patients

CONTACTS AND LOCATIONS:
Locations (1):
- Lifebrain Cerba Healthcare laboratory network, Guidonia, Roma, Italy